CLINICAL TRIAL: NCT03181932
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Study of AeroVanc for the Treatment of Persistent Methicillin-resistant Staphylococcus Aureus Lung Infection in Cystic Fibrosis Patients
Brief Title: AeroVanc in the Treatment of Methicillin-resistant Staphylococcus Aureus Infection in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAV005-04
Record Dates: First submitted 2017-06-01; First posted 2017-06-09 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: MRSA; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blind vancomycin inhalation powder (Experimental): Vancomycin inhalation powder 30 mg is administered twice daily (BID) during the 24-week double-blind period (Period 1) by inhalation during three dosing cycles, each cycle being 28 days of treatment followed by 28 days of observation.
  Interventions: Drug: Vancomycin inhalation powder
- Double-blind placebo inhalation powder (Placebo Comparator): Matching placebo is administered BID during the 24-week double-blind period (Period 1) by inhalation during three dosing cycles, each cycle being 28 days of treatment followed by 28 days of observation.
  Interventions: Drug: Placebo inhalation powder
- Open-label vancomycin inhalation powder (Experimental): In the 24-week Period 2, all participants receive AeroVanc 30 mg BID by inhalation during three dosing cycles, each cycle being 28 days of treatment followed by 28 days of observation.
  Interventions: Drug: Vancomycin inhalation powder

INTERVENTIONS:
Drug: Vancomycin inhalation powder — 100 participants are to be treated with double-blind vancomycin inhalation powder (75 subjects ≤21 years old, 25 subjects >21 years old) for 24 weeks during Period 1.
  Other Names: AeroVanc
  Arms: Double-blind vancomycin inhalation powder
Drug: Placebo inhalation powder — 100 participants are to be treated with double-blind placebo (75 subjects ≤21 years old, 25 subjects >21 years old) for 24 weeks during Period 1.
  Arms: Double-blind placebo inhalation powder
Drug: Vancomycin inhalation powder — In the 24-week Period 2, all participants are to be treated with open-label vancomycin inhalation powder.
  Other Names: AeroVanc
  Arms: Open-label vancomycin inhalation powder

SUMMARY:
This is a multi-center, randomized phase III study to evaluate the clinical effectiveness of AeroVanc in persistent methicillin-resistant Staphylococcus aureus (MRSA) infection in patients with cystic fibrosis (CF).

DETAILED DESCRIPTION:
This is a phase III, randomized, multicenter, double-blind, placebo-controlled, parallel-group study to examine the safety and efficacy of AeroVanc in the treatment of persistent MRSA lung infection in patients diagnosed with CF. After the Screening period to confirm study eligibility, participants are randomly assigned in a blinded fashion to receive either AeroVanc 30 mg twice daily (BID), or placebo BID (1:1 active to placebo) by inhalation for 24 weeks or 3 dosing cycles (Period 1). Upon completion of Period 1, participants receive open-label AeroVanc 30 mg BID for an additional 24 weeks or 3 dosing cycles (Period 2), to evaluate long-term safety of AeroVanc. A dosing cycle is defined as 28 days of treatment followed by 28 days of observation.

Participants on a 28-day cyclical on/off anti-Pseudomonal antibiotic regimen enter the Screening period at a time such that the Baseline visit coincide with the end of their anti-Pseudomonas antibiotic cycle. Study drug is thereby administered during the off-cycle, and participants can then resume anti-Pseudomonal therapy during the 28-day observation period. Participants continuing alternating anti-Pseudomonal therapy can continue their treatment during the study drug administration, and observation period.

The primary and secondary analyses are conducted in participants ≤21 years old. Subjects >21 years old are analyzed separately as supportive analyses.

ELIGIBILITY:
Inclusion criteria

1. Participants ≥6 years of age at time of informed consent form or assent form signing.
2. Confirmed diagnosis of CF, determined by having clinical features consistent with the CF phenotype, plus one of the following:

   1. Positive sweat chloride test (value ≥60 milliequivalent/L),
   2. Genotype with 2 mutations consistent with CF (i.e., a mutation in each of the cystic fibrosis transmembrane conductance regulator genes).
3. Positive sputum culture or a throat swab culture for MRSA at Screening.
4. In addition to the Screening sample, have at least 2 prior sputum or throat swab cultures positive for MRSA, of which at least 1 sample is >6 months prior to Screening. At least 50% of all MRSA cultures (sputum or throat swab culture) collected from the time of the first positive culture (in the previous 1 year) must have tested positive for MRSA. (Note: Screening sample may count towards 50% positive count)
5. FEV1 ≥30% and ≤90% of predicted that is normal for age, gender, race, and height, using the Global Lung Function Initiative equation.
6. At least 1 episode of acute pulmonary infection treated with non-maintenance antibiotics within 12 months prior to the Baseline visit (initiation of treatment with intermittent inhaled anti-Pseudomonal therapy will not qualify as treatment with non-maintenance antibiotics).
7. If female of childbearing potential, an acceptable method of contraception must be used during the study and must be combined with a negative pregnancy test obtained during Screening; sexually active male subjects of reproductive potential who are non-sterile (i.e., male who has not been sterilized by vasectomy for at least 6 months, and were not diagnosed with infertility through demonstration of azoospermia in a semen sample and/or absence of vas deferens through ultrasound) must be willing to use a barrier method of contraception, or their female partner must use an acceptable method of contraception, during the study.

   For purposes of this study, the Sponsor defines "acceptable methods of contraception" as:
   1. Oral birth control pills administered for at least 1 monthly cycle prior to administration of the study drug.
   2. A synthetic progestin implanted rod (eg, Implanon®) for at least 1 monthly cycle prior to the study drug administration but not beyond the 4th successive year following insertion.
   3. Intrauterine devices, inserted by a qualified clinician for at least 1 monthly cycle prior to study drug administration.
   4. Medroxyprogesterone acetate (eg, Depo-Provera®) administered for a minimum of 1 monthly cycle prior to administration of the study drug and continuing through 1 month following study completion.
   5. Hysterectomy or surgical sterilization.
   6. Abstinence.
   7. Double barrier method (diaphragm with spermicidal gel or condoms with contraceptive foam).

   Note: For subjects prescribed Orkambi: Orkambi may substantially decrease hormonal contraceptive exposure, reducing the effectiveness and increasing the incidence of menstruation-associated adverse reactions. Hormonal contraceptives, including oral, injectable, transdermal, and implantable, should not be relied upon as an effective method of contraception when co-administered with Orkambi.
8. Able and willing to comply with the protocol, including availability for all scheduled study visits and able to perform all techniques necessary to use the AeroVanc inhaler and measure lung function.
9. Agree not to smoke during any part of the clinical trial (Screening visit through end of study).
10. Participants with a Pseudomonas aeruginosa co-infection must either be stable on a regular suppression regimen of inhaled antibiotics or must be, in the opinion of the Investigator, stable despite the lack of such treatment.

Exclusion criteria

1. Use of anti-MRSA treatments prescribed as maintenance therapy (intravenous [IV] or inhaled treatment within 28 days; oral treatment within 14 days) prior to the Baseline visit.
2. Use of non-maintenance antibiotic for pulmonary infection or extrapulmonary MRSA infection (IV or inhaled antibiotic within 28 days; oral antibiotic within 14 days) prior to the Baseline visit.
3. History of previous allergies or sensitivity to vancomycin, or other component(s) of the study drug or placebo except for a history of red-man syndrome.
4. Inability to tolerate inhaled products.
5. First time sputum culture or throat swab culture yielding Burkholderia cepacia, or nontuberculous Mycobacteria in the previous 6 months to Screening.
6. History of lung or other solid organ transplantation or currently on the list to receive lung or other solid organ transplantation.
7. Resistance to vancomycin at Screening (vancomycin resistant Staphylococcus aureus, or vancomycin intermediate resistant Staphylococcus aureus, with minimum inhibitory concentration ≥8 μg/mL).
8. Oral corticosteroids in doses exceeding 10 mg prednisone per day or 20 mg prednisone every other day, or equipotent doses of other corticosteroids.
9. Changes in antimicrobial, bronchodilator, anti-inflammatory or corticosteroid medications within 14 days, or changes in cystic fibrosis transmembrane conductance modulators within 28 days, prior to the Baseline visit.
10. Abnormal laboratory findings or other findings or medical history at Screening that, in the Investigator's opinion, would compromise the safety of the subject or the quality of the study data.
11. Inability to tolerate inhalation of a short acting beta2 agonist
12. Oxygen saturation <90% at Screening.
13. Changes in physiotherapy technique or physiotherapy scheduled within 1 week of the Baseline visit.
14. Administration of any investigational drug or device within 4 weeks prior to the Screening visit and during the study
15. Female with positive pregnancy test result during Screening, pregnant (or intends to become pregnant), lactating or intends to breastfeed during the study.
16. Renal insufficiency, defined as creatinine clearance <50 mL/min using the Cockcroft-Gault equation for adults or Schwartz equation for children at the Screening visit.
17. Abnormal liver function, defined as ≥4x upper limit of normal of serum aspartate aminotransferase or serum alanine aminotransferase, or known cirrhosis at Screening.
18. Diagnosed with clinically significant hearing loss.
19. History of positive result for human immunodeficiency virus, hepatitis B virus or hepatitis C virus.
20. Planned hospitalizations for prophylaxis antibiotic treatment within 28 days prior to Baseline visit or during the double-blind period (Period 1).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flume, MD, Principal Investigator — Medical University of South Carolina
Locations (71):
- United States (69):
  - Pulmonary Associates of Mobile, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Miller Childrens Hospital MemorialCare Health System Pediatric Pulmonology, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Southern California Keck Medical Center of USC, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health Adult Cystic Fibrosis Center, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Pediatrics, Gainesville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Nemours Childrens Specialty Care, Jacksonville, Florida
  - University of Miami Bachelor Children's Hospital, Miami, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Arnold Palmer Hospital Pulmonary and Sleep Medical Institute Orlando Health, Inc, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Specialty Care, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Health Care of Atlanta at Scottish Rite, Atlanta, Georgia
  - Augusta Univ Cystic Fibrosis Center, Augusta, Georgia
  - Chicago CF Care Specialists, Glenview, Illinois
  - NorthSurburban Pulmonary Specialists, Morton Grove, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Iowa Department of Pediatrics, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Via Christi Health Systems CF Clinic, Wichita, Kansas
  - University of Louisville Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Maine Medical Partners Pediatric Specialty Care, Portland, Maine
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University (HUH), Detroit, Michigan
  - Children's Mercy, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital /Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Pediatric/Pulmonary, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Northwell Health, Div of Pulmonary, Critical Care & Sleep Medicine, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Levine Children's Hospital - Atrium Health, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Toledo Children's Hospital CF Center, Toledo, Ohio
  - University of Oklahoma Health Science Center - Pediatric Pulmonary & CF Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMCU, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sanford Childrens Specialty Clinic, Sioux Falls, South Dakota
  - UTHSC Lebonheur Children's Hospital, Memphis, Tennessee
  - Austin Children's Chest Associates, Austin, Texas
  - Children's Medical Center Cystic Fibrosis Clinic, Dallas, Texas
  - Cook Children Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University Vermont Medical Center Vermont Lung Center, Colchester, Vermont
  - University of Virginia Health System, Cystic Fibrosis Center, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Medical Research Center, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo DK, Muhlebach MS, Smyth AR. Interventions for the eradication of meticillin-resistant Staphylococcus aureus (MRSA) in people with cystic fibrosis. Cochrane Database Syst Rev. 2022 Dec 13;12(12):CD009650. doi: 10.1002/14651858.CD009650.pub5. PMID 36511181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 76 sites in Canada (2 clinics) and US (74 clinics) enrolled participants in the trial. First participant was enrolled on 20 September 2017 and last subject completed the study on 15 January 2021.
Pre-assignment Details: A total of 353 participants were screened, and 188 were randomized in Period 1. In total, 165 participants were screen failures and the reasons for screen failure were ineligibility (n=157), exacerbation (n=6), lost to follow-up (n=1) and other reason (n=1).
Period: Period 1 (Double-blind Period)
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Started (The number of started participants include both age groups (participants 6-21 years and >21 years). The primary efficacy population was the 6-21 years age group. All Outcome Results are presented for the primary age group. The Baseline Characteristics and Safety Results are presented for all participants.) | 90 | 98
Completed | 79 | 85
Not Completed | 11 | 13
Not completed — Adverse Event | 5 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 5 | 9
Period: Period 2 (Open-label Period)
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Started (The numbers refer to the treatment that the participants received during Period 1. 6 participants (4 in the vancomycin group and 2 in the placebo group) who completed Period 1 decided not to participate in Period 2.) | 75 | 83
Completed | 67 | 70
Not Completed | 8 | 13
Not completed — Adverse Event | 1 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Reason missing | 2 | 0

BASELINE CHARACTERISTICS:
Population: The number of baseline participants include both age groups (participants 6-21 years and >21 years).
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder | Total
Number analyzed (Participants) | 90 | 98 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (12.52) | 18.2 (8.70) | 19.2 (10.71)
Age, Customized [Count of Participants; unit: Participants]
  6-21 years | 64 | 69 | 133
  >21 years | 26 | 29 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 95
  Male | 45 | 48 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 86 | 92 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 85 | 94 | 179
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Pseudomonas Aeruginosa Infection Present at Screening (Yes/No?) [Count of Participants; unit: Participants]
  Yes | 51 | 45 | 96
  No | 39 | 53 | 92
Number of Pulmonary Infections in the Previous Year [Mean (Standard Deviation); unit: infections] | 2.6 (1.53) | 2.6 (1.44) | 2.6 (1.48)
Baseline Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted [Mean (Standard Deviation); unit: percent predicted] | 65.25 (16.193) | 66.32 (16.939) | 65.81 (16.550)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted
Description: The mean absolute change from baseline in FEV1 percent predicted was analyzed sequentially at Week 4 (end of Cycle 1), Week 12 (end of Cycle 2) and at Week 20 (end of Cycle 3).
Time Frame: Baseline and Week 4, 12 and 20
Population: Intention-to-treat (ITT) population (defined as all randomized participants). Participants were analyzed according to randomized treatment. The ITT population was also split out by age (≤21 years, >21 years). The population of participants ≤21 years was used for all main analyses of efficacy endpoints.
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 64 | 69
Percent predicted
  Week 4 | 2.39 (8.078) | 1.18 (8.581)
  Week 12 | 1.52 (8.414) | 0.13 (8.056)
  Week 20 | 1.61 (9.967) | -1.94 (8.924)
Statistical Analysis 1: Comparison: Double-blind Vancomycin Inhalation Powder vs Double-blind Placebo Inhalation Powder; Based on previous experience, a sample size of 45 participants per arm would provide 89% power to detect a statistically significant difference at alpha level of 0.05. To account for potential dropouts and/or smaller effect size in a 3-cycle trial, a sample size of 75 participants per arm was to be enrolled in the primary analysis population, which if all completed would provide 90% power to detect a difference of 3.4% at 20 weeks assuming the same standard deviation of 6.3%; Test type: Superiority — The primary efficacy endpoint was tested sequentially at Week 4 (end of Cycle 1), Week 12 (end of Cycle 2) and at Week 20 (end of Cycle 3). If a statistically significant difference was observed in favor of vancomycin inhalation powder compared to placebo after Cycle 1, then the mean change in the FEV1 percent predicted during Cycle 2 was to be tested. Similarly, if the effect after Cycle 2 was statistically significant, then the analysis of Baseline to end of Cycle 3 was to be tested; p = 0.325, Mixed Models Analysis; Least square mean difference = 1.4, 95% CI 2-sided [-1.4 to 4.1]

2. Secondary Outcome: Frequency of Pulmonary Exacerbations
Description: The number of pulmonary exacerbations during Period 1 adjusted for the length of follow-up.
Time Frame: Week 20
Population: ITT population (6-21 years).
Measure: Mean (Standard Deviation); unit: exacerbations
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 64 | 69
exacerbations | 0.9 (1.03) | 0.9 (1.02)

3. Secondary Outcome: Time to First Pulmonary Exacerbation
Description: Time to first pulmonary exacerbation requiring use of another antibiotic medication (oral, IV, and/or inhaled). The Outcome Measure Data presented are the median percentiles and 95% confidence intervals from Kaplan-Meier estimates.
Time Frame: Week 20
Population: ITT population (6-21 years).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 64 | 69
days | 38 [18 to 49] | 48 [29 to 59]

4. Secondary Outcome: Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Scores
Description: The CFQ-R was administered every two weeks using a hand-held e-Diary. CFQ-R scores range between 0 and 100, where higher scores indicate a better outcome. The CFQ-R measures functioning in a variety of domains, including Physical Functioning, Vitality, Health Perceptions, Respiratory Symptoms, Treatment Burden, Role Functioning, Emotional Functioning and Social Functioning. The Outcome Measure Data presented are the Respiratory Symptoms Scores.
Time Frame: Baseline and Week 4, 12, and 20
Population: ITT population (6-21 years).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 64 | 69
score on a scale
  Week 4 | 8.4 [4.2 to 12.7] | 3.0 [-1.0 to 7.0]
  Week 12 | 6.0 [1.4 to 10.6] | 4.3 [-0.2 to 8.9]
  Week 20 | 4.6 [-0.8 to 10.1] | 6.3 [1.2 to 11.4]

5. Secondary Outcome: Change From Baseline in Cystic Fibrosis Respiratory Symptom Diary-Chronic Respiratory Symptom Score (CFRSD-CRISS) Scores
Description: The CFRSD-CRISS was administered every two weeks using a hand-held e-Diary. Scores range between 0 and 100, where higher scores indicate a worse outcome.
Time Frame: Baseline and Week 4, 12 and 20
Population: ITT population (6-21 years).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 64 | 69
score on a scale
  Week 4 | -3.2 [-7.3 to 0.9] | -5.1 [-9.1 to -1.1]
  Week 12 | -4.7 [-10.1 to 0.6] | -8.0 [-13.3 to -2.8]
  Week 20 | -7.3 [-12.5 to -2.0] | -5.3 [-10.3 to -0.4]

6. Secondary Outcome: Relative Change in FEV1 Percent Predicted
Description: The mean relative change from Baseline in FEV1 percent predicted
Time Frame: Baseline and Week 4, 12 and 20
Population: ITT population (6-21 years).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 64 | 69
percent predicted
  Week 4 | 2.9 [-1.0 to 6.8] | 1.5 [-2.1 to 5.1]
  Week 12 | 1.2 [-2.8 to 5.2] | -0.3 [-4.1 to 3.5]
  Week 20 | 1.7 [-2.7 to 6.1] | -2.2 [-6.4 to 2.0]

7. Secondary Outcome: Number of Successful Response Cycles
Description: The number of successful response cycles a participant achieves over Period 1. A response in a cycle is defined by at least a 5 % relative improvement in FEV1 percent predicted at the end of each the respective cycle.
Time Frame: Week 20
Population: ITT population (6-21 years).
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 62 | 66
Participants
  0 successful response cycles | 20 | 24
  1 successful response cycle | 18 | 27
  2 successful response cycles | 15 | 9
  3 successful response cycles | 9 | 6

8. Secondary Outcome: Area Under the FEV1-time Profile
Description: The mean treatment difference in FEV1 across all post-baseline visits
Time Frame: Week 20
Population: ITT population (6-21 years).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted*hour/liter
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder
Number analyzed (Participants) | 64 | 69
percent predicted*hour/liter | 609.7 [520.8 to 698.7] | 583.1 [499.8 to 666.5]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were assessed on or after the first dose of trial drug to 28 days after last dose. For all safety analyses, a single set of results was produced including all participants (6-21 and >21 years combined). For the double-blind Period 1, AE data are presented for the vancomycin and placebo groups whereas for the open-label Period 2, AE data for only one combined group is presented.
Groups:
- Double-blind Vancomycin Inhalation Powder: Vancomycin inhalation powder 30 mg is administered twice daily (BID) during the 24-week double-blind period (Period 1) by inhalation during three dosing cycles, each cycle being 28 days of treatment followed by 28 days of observation.
  Vancomycin inhalation powder: 100 participants are to be treated with double-blind vancomycin inhalation powder (75 participants ≤21 years old, 25 participants >21 years old) for 24 weeks during Period 1.
- Double-blind Placebo Inhalation Powder: Matching placebo is administered BID during the 24-week double-blind period (Period 1) by inhalation during three dosing cycles, each cycle being 28 days of treatment followed by 28 days of observation.
  Placebo inhalation powder: 100 participants are to be treated with double-blind placebo (75 participants ≤21 years old, 25 participants >21 years old) for 24 weeks during Period 1.
- Open-label Vancomycin Inhalation Powder: In the 24-week Period 2, all participants receive vancomycin inhalation powder 30 mg BID by inhalation during three dosing cycles, each cycle being 28 days of treatment followed by 28 days of observation.
  Vancomycin inhalation powder: In the 24-week Period 2, all participants are to be treated with open-label vancomycin inhalation powder.
Arm/Group | Double-blind Vancomycin Inhalation Powder | Double-blind Placebo Inhalation Powder | Open-label Vancomycin Inhalation Powder
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/98 | 0/158
Serious Adverse Events (participants affected / at risk) | 24/90 | 35/98 | 50/158
Other Adverse Events (participants affected / at risk) | 85/90 | 93/98 | 139/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Vancomycin Inhalation Powder (N=90) | Double-blind Placebo Inhalation Powder (N=98) | Open-label Vancomycin Inhalation Powder (N=158)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 19 (24) | 29 (33) | 38 (43)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 2 (3) | 3 (3) | 3 (3)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Systemic viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (6) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Vancomycin Inhalation Powder (N=90) | Double-blind Placebo Inhalation Powder (N=98) | Open-label Vancomycin Inhalation Powder (N=158)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 51 (109) | 59 (116) | 78 (140)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 4 (5) | 12 (15)
Pneumonia (Infections and infestations) | 5 (7) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 5 (5) | 6 (6) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (62) | 36 (53) | 40 (50)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 10 (15) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (16) | 9 (9)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 7 (10) | 9 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (9) | 8 (9)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (8) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5) | 8 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (10) | 11 (14) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (6) | 7 (13) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 10 (11) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (11) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 7 (9) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 7 (8) | 0 (0)
Forced expiratory volume decreased (Investigations) | 1 (1) | 6 (6) | 0 (0)
Glucose urine present (Investigations) | 2 (2) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 11 (12) | 8 (10) | 8 (9)
Chest discomfort (General disorders) | 9 (10) | 8 (8) | 0 (0)
Fatigue (General disorders) | 3 (5) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 9 (13) | 12 (14) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
A total of 200 participants were to be randomized. Consequent to the outbreak of COVID-19, the recruitment was stopped prematurely when 188 participants had been randomized.

The CFQ-R and CFRSD-CRISS were administered every two weeks using a hand-held e-Diary. The e-Diary had not been activated at the baseline visit for 39 participants. For these participants, missing baseline measurements were imputed with the population median baseline value for inferential analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03181932/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03181932/SAP_001.pdf